CLINICAL TRIAL: NCT00675532
Title: Testing a Primary Care Model for the Treatment of Opioid Dependence Using Long-acting Injectable Naltrexone (Vivitrol).
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, David Fiellin, Associate Professor of Internal Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yale HIC #0708002942
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Drug Dependence
Keywords: Opioids, vivitrol, naltrexone, primary care
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Primary Care Counseling
  Interventions: Behavioral: Primary Care Counseling
- 2 (Experimental): Cognitive-behavioral psychotherapy (CBT)
  Interventions: Behavioral: Cognitive-behavioral psychotherapy

INTERVENTIONS:
Behavioral: Primary Care Counseling — Subjects in this condition will attend bi-weekly 15 minute sessions with the study nurse for primary care counseling which is a brief manual-guided, medically focused counseling approach to the treatment of opioid dependent individuals seen in primary care settings. The brief counseling sessions involve repeated support for and monitoring of medication compliance, and the provision of advice regarding established methods for coping with psychological and social factors that lead to drug use.
  Arms: 1
Behavioral: Cognitive-behavioral psychotherapy — Subjects in the CBT condition will participate in bi-weekly 50-minute-long individualized cognitive-behavioral psychotherapy sessions with a CBT trained clinician. The general purpose of the therapy is to: (1) acquire information about important concepts and aspects of recovery from opioid addiction; (2) increase self-awareness of specific problems and issues in relation to addiction and recovery, and (3) learn new coping skills to deal with problems contributing to or resulting from the addiction and to improve overall psychosocial functioning. The primary focus of this approach is to provide patients with frequent supportive contact and to teach cognitive-behavioral relapse prevention skills.
  Arms: 2

SUMMARY:
In opioid dependent patients treated with long-acting injectable naltrexone (Vivitrol ®), we will compare the efficacy of a primary care model of counseling (Condition 1) versus individualized cognitive-behavioral psychotherapy (Condition 2) for the treatment of opioid dependence. Treatment will last 12 weeks, and participants will be given 380mg of naltrexone per injection (3 injections in total; each lasting 4 weeks). Primary outcomes will be 1) percent of opioid negative urines and 2) treatment compliance as measured by attendance and time in treatment. Secondary outcomes are opiate craving, opiate withdrawal symptoms, perceived stress scores, severity of addiction problems, and patient satisfaction. Findings will elucidate whether injectable, long-acting naltrexone would be safe and effective in a primary care setting where medication would be administered in the absence of traditional cognitive-behavioral psychotherapy and indicate whether cognitive-behavioral psychotherapy adds to treatment effects above and beyond primary care counseling. If positive, this small controlled study will provide effect size estimates for a larger trial to assess Vivitrol ® in a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals, ages 18 and above, meeting current diagnostic and statistical manual (DSM-IV) criteria for opioid dependence.
* Subject has voluntarily given informed consent and signed the informed consent document.
* Able to read English and complete study evaluations.

Exclusion Criteria:

* Regular use of benzodiazepines.
* Psychotic or otherwise severely psychiatrically disabled (i.e., suicidal, homicidal, current mania);
* Significant underlying medical conditions such as cerebral, renal, thyroid or cardiac pathology which in the opinion of study physician would preclude patient from fully cooperating or be of potential harm during the course of the study;
* Abstinent from opiates for more than four weeks prior to naltrexone initiation.
* Medical problems that would preclude naltrexone treatment, such as laboratory evidence of significant hepato-cellular injury as evidenced by abnormal liver enzyme tests including SGOT and SGPT (> three times normal) or elevated bilirubin levels), and a history of cirrhosis.
* Women who are pregnant, nursing or refuse to use a reliable form of birth control (as assessed by pregnancy tests during initial evaluation for naltrexone, and every two weeks during the course of the study).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Primary outcomes will be 1) percent of opioid negative urines and 2) treatment compliance as measured by attendance and time in treatment. | 12 weeks

SECONDARY OUTCOMES:
Secondary outcomes are opiate craving, opiate withdrawal symptoms, perceived stress scores, severity of addiction problems, and patient satisfaction. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Fiellin, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Primary Care Center, New Haven, Connecticut, United States